CLINICAL TRIAL: NCT02156180
Title: A Prospective Cohort Study to Determine Specific Volatile Organic Compounds Present in Breath Samples of Patients With Oral Cavity or Oropharyngeal Squamous Cell Carcinoma Using Gas Chromotography-mass Spectrometry
Brief Title: Identification of Breath Biomarkers in Head and Neck Squamous Cell Carcinoma
Status: Suspended | Type: Observational
Why Stopped: Awaiting funding to facilitate selected-ion flow-tube mass spectrometry (SIFT/MS)
Sponsor: Queensland Centre of Excellence for Head and Neck Cancer (Other)
Collaborators: Princess Alexandra Hospital, Brisbane, Australia (Other); Queensland Health Forensic and Scientific Services (Unknown)
Responsible Party: Sponsor
Other Study IDs: HREC14QPAH10
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Oral Cavity Squamous Cell Carcinoma; Oropharyngeal Squamous Cell Carcinoma
Keywords: exhaled breath; volatile organic compounds; surgery; chemotherapy; radiotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Early stage oral cavity / oropharyngeal cancer: Exhaled breath

SUMMARY:
In this study the Investigators aim to determine specific volatile compounds present in breath samples of patients with oral cavity or oropharyngeal squamous cell carcinoma before and after tumour resection or before and after chemotherapy +/- radiotherapy using gas chromotography-mass spectrometry. The Investigators hypothesize that study participants with a tumour will display a distinct set of volatile organic compounds than can serve as potential cancer biomarkers.

DETAILED DESCRIPTION:
Head and neck cancer diagnosis is devastating as it frequently disrupts one's ability to communicate, swallow and breathe. Each year, physicians diagnose approximately 650,000 cases of head and neck cancer worldwide. Many people with head and neck cancer have their cancer detected late, and this can result in a poor clinical outcome. One strategy to improve the clinical outcomes for people with a head and neck cancer is to develop a non-invasive screening assay using breath biomarkers. Such a diagnostic tool will identify at-risk individuals early, and potentially offer improved and cost-effective treatment.

The idea of using human breath samples to detect cancer began with the observation that dogs can be trained to "sniff out" certain types of cancers from urine and blood. Since then the presence of various volatile organic compounds from many types of cancers, including: lung, skin, breast, prostate, and bladder have been characterized. These studies are ongoing, but promise to revolutionize the way physicians screen cancer in the future.

In this pilot study, the Investigators aim to determine specific volatile organic compounds present in breath samples of patients with oral cavity or oropharyngeal cancer before and after tumor resection, or before and after definitive chemotherapy/radiotherapy. As head and neck cancer can result in significant functional deficit, early detection is the key to improving clinical outcome. Much anecdotal evidence exists for the presence of distinct odor emissions from the tumor bed of head and neck cancer patients. Therefore, the identification of specific volatile organic compound to head and neck cancer will undoubtedly lead to a novel, cost-effective screening strategy for early detection of head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years
* Clinical diagnosis of oral cavity or oropharyngeal squamous cell carcinoma

Exclusion Criteria:

* Evidence of metastatic disease
* Previous treatment of this cancer with surgery, chemotherapy or radiotherapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who attend the Head and Neck Cancer Clinic at the Princess Alexandra Hospital, Brisbane, Australia
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Presence of volatile organic compounds in breath samples if patients with oral cavity or oropharyngeal squamous cell carcinoma | Approximately 1-4 months
  Breath samples of patients with oral cavity or oropharyngeal squamous cell carcinoma will be compared before treatment - surgery or radiotherapy/chemotherapy, and then one month after completion of treatment - surgery or radiotherapy/chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jae Lim, Dr, Principal Investigator — Princess Alexandra Hospital; Ben Panizza, Assoc Prof, Principal Investigator — Princess Alexandra Hospital; Vince Alberts, Mr, Principal Investigator — Queensland Health Forensic and Scientific Services; Jeff Herse, Mr, Principal Investigator — Queensland Health Forensic and Scientific Services; David Pass, Mr, Principal Investigator — Queensland Health Forensic and Scientific Services; Nigel Brown, Dr, Principal Investigator — Princess Alexandra Hospital
Locations (1):
- Princess Alexandra Hospital, Brisbane, Queensland, Australia

REFERENCES:
- [Background] Willis CM, Church SM, Guest CM, Cook WA, McCarthy N, Bransbury AJ, Church MR, Church JC. Olfactory detection of human bladder cancer by dogs: proof of principle study. BMJ. 2004 Sep 25;329(7468):712. doi: 10.1136/bmj.329.7468.712. PMID 15388612
- [Background] Chan HP, Lewis C, Thomas PS. Exhaled breath analysis: novel approach for early detection of lung cancer. Lung Cancer. 2009 Feb;63(2):164-8. doi: 10.1016/j.lungcan.2008.05.020. Epub 2008 Jul 2. PMID 18599152
- [Background] Lippi G. Re: Jean-Nicolas Cornu,Geraldine Cancel-Tassin, Valerie Ondet, et Al. Olfactory detection of prostate cancer by dogs sniffing urine: a step forward in early diagnosis. Eur urol 2011; 59: 197-201. Eur Urol. 2011 Oct;60(4):e29; author reply e30. doi: 10.1016/j.eururo.2011.06.030. Epub 2011 Jun 22. No abstract available. PMID 21726935
- [Background] Badjagbo K. Exhaled breath analysis for early cancer detection: principle and progress in direct mass spectrometry techniques. Clin Chem Lab Med. 2012 Nov;50(11):1893-1902. doi: 10.1515/cclm-2012-0208. PMID 22718640
- [Background] Dobrossy L. Epidemiology of head and neck cancer: magnitude of the problem. Cancer Metastasis Rev. 2005 Jan;24(1):9-17. doi: 10.1007/s10555-005-5044-4. PMID 15785869